CLINICAL TRIAL: NCT04252274
Title: Efficacy and Safety of Darunavir and Cobicistat for Treatment of COVID-19
Acronym: DC-COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC-COVID-19
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia, Pneumocystis; Coronavirus
Keywords: Pneumonia; COVID-19; Darunavir; Cobicistat
MeSH Terms: conditions — Pneumonia, Pneumocystis; Coronavirus Infections; Pneumonia; COVID-19 | interventions — cobicistat mixture with darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darunavir, Cobicistat and conventional treatments (Experimental): After randomization, subjects take darunavir and cobicistat one tablet per day for 5 days, also take conventional treatments.
  Interventions: Drug: Darunavir and Cobicistat
- Conventional treatments (No Intervention): After randomization, subjects take conventional treatments without darunavir and cobicistat.

INTERVENTIONS:
Drug: Darunavir and Cobicistat — Subjects take darunavir and cobicistat one tablet per day for 5 days, also take conventional treatments
  Arms: Darunavir, Cobicistat and conventional treatments

SUMMARY:
The study aims to evaluate the efficacy and safety of darunavir and cobistastat in the treatment of COVID-19 pneumonia

DETAILED DESCRIPTION:
There is no vaccine or antiviral treatment for human coronavirus, so this study aims to evaluate the efficacy and safety of darunavir and cobistastat in the treatment of COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* The participants were diagnosed as COVID-19 pneumonia, according to the notice on printing and distributing the diagnosis and treatment plan of pneumonia with new coronavirus infection (trial version 4 or update version) made by National Health Commission of the People's Republic of China.
* Written the informed consent

Exclusion Criteria:

* Hypersensitivity to darunavir, cobicistat, or any excipients
* Patients with severe liver injury (Child-Pugh Class C)
* Concomitant medications that are highly dependent on CYP3A clearance, and the elevated plasma concentrations are associated with serious or life-threatening events.
* Subjects were considered to be unable to complete the study, or not suitable for the study by researchers

Exit criteria:

* Subjects asked to withdraw the study
* Subject will benefit if withdraw according to researchers' suggestions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 7 | 7 days after randomization

SECONDARY OUTCOMES:
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 3 | 3 days after randomization
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 5 | 5 days after randomization
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 14 days after randomization
The critical illness rate of subjects at weeks 2 | 14 days after randomization
  The diagnosis of critical illness case was based on the notice on printing and distributing the diagnosis and treatment plan of pneumonia with new coronavirus infection (trial version 4) made by National Health Commission of the People's Republic of China.
The mortality rate of subjects at weeks 2 | 14 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen J, Xia L, Liu L, Xu Q, Ling Y, Huang D, Huang W, Song S, Xu S, Shen Y, Lu H. Antiviral Activity and Safety of Darunavir/Cobicistat for the Treatment of COVID-19. Open Forum Infect Dis. 2020 Jun 21;7(7):ofaa241. doi: 10.1093/ofid/ofaa241. eCollection 2020 Jul. PMID 32671131